CLINICAL TRIAL: NCT05978440
Title: Clinical and Laboratory Evaluation of Cad-cam Restorations Fabricated From Digital Impression Under Rubber Dam Isolation (Randomized Clinical Trial & In-vitro Study)
Brief Title: This Trial Will Evaluate the Clinical Performance of Onlay Restorations Fabricated Using Rubber Dam Scanning Techniques.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0682-05/2023 IRB 00010556; IRB 00010556 (Registry Identifier: ethical approval number)
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Inlays

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scanning without rubber dam (Active Comparator): After the onlay preparation, standard digital impression will be recorded for the working quadrant using the IOS without applying the rubber dam. Then the opposing quadrant will be scanned in addition to interocclusal bite registration.
  Interventions: Procedure: onlay preparation
- Scanning under rubber dam with cut technique (Experimental): In this group a pre-operative scan will be already taken before the preparation for the working arch, opposing arch and the interocclusal bite registration. Then using the "Cut" feature in the software of the IOS to cut the area of the working tooth. After the preparation, rubber dam will be applied on the working quadrant and then rescan the prepared tooth.
  Interventions: Procedure: onlay preparation
- Scanning under rubber dam with new lock technique (Experimental): After the onlay preparation, the rubber dam will be applied to the working quadrant. Digital impression will be taken using the IOS. After that using the "lock" feature in the software of the scanner, all the preparation area and margins will be locked. Rubber dam will be removed, and scanning will be completed for the whole quadrant and opposing arch in addition to interocclusal bite registration.
  Interventions: Procedure: onlay preparation

INTERVENTIONS:
Procedure: onlay preparation — CAD-CAM onlay restorations will be fabricated using rubber dam scanning techniques and evaluated clinically up to 12 months

SUMMARY:
The purpose of this study will be to evaluate the clinical performance of CAD-CAM onlay restorations fabricated using rubber dam scanning techniques up to 12 months and laboratory investigation of their marginal fit.

DETAILED DESCRIPTION:
A total of 54 molars will be prepared for CAD-CAM onlay restorations. The preparations will be divided into three groups according to the technique of scanning. Group I: 18 preparations will be scanned without rubber dam using standard technique, group II: 18 preparations will be scanned under rubber dam isolation using cut technique, and group III: 18 preparations will be scanned under rubber dam isolation using lock technique. Final restorations will be milled, checked and cemented, then will be evaluated using the modified FDI criteria at baseline, three months, six months, and one year.

Thirty resin dies will be 3D printed after scanning of a first molar tooth prepared for onlay. The dies will be scanned after they fit in a typodont and grouped with the same technique (n=10 per group). The digital scans will be superimposed using a 3D best-fit alignment method and 3D deviation will be calculated for each group itself and to the other groups. The marginal fit of the restorations produced will be checked using two methods: Triple scan and measuring the cement thickness after cementation and sectioning of the samples.

All data will be collected, and statistically analyzed using suitable tests.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult patients (18-45 years old).
2. Patients in need of class II (OM or OD) caries in molar teeth with initial, moderate or extensive stage according to the staging of caries lesions in The International Caries Detection and Assessment system (ICDASTM codes 2 to 6) (32,33).
3. Presence of proximal caries in digital x-ray with score 2 to 4 according to the ICDAS/ICCMS™ radiographic scoring system(32,33).
4. Vital teeth with absence of clinical signs and symptoms of periapical pathology.
5. Patient Ability to tolerate Rubber Dam applications.
6. Patients who will agree to attend regular check-ups.

Exclusion Criteria:

1. Bad oral hygiene (Grade 3)(34).
2. Non- vital teeth or endodontically treated teeth.
3. Severe Periodontal problems (pockets ≥6mm).
4. Patients with para-functional habits (e.g., Bruxism, attrition, wear facets)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical performance of CAD-CAM onlay restorations fabricated using rubber dam scanning. | 12 months
  Restorations will be evaluated according to three main domains: (40)
  1. Functional (domain F): fracture of material and retention(F1), marginal adaptation(F2), proximal contact point(F3), Form and contour(F4), and Occlusion and wear(F5).
  2. Biological (domain B): Caries at restoration margins(B1), dental hard tissue defects at restoration margin(B2), postoperative hypersensitivity/pulp status(B3).
  3. Aesthetics (domain A): Surface luster and surface texture(A1), Marginal staining(A2), Color match(A3).

CONTACTS AND LOCATIONS:
Overall Officials: hossam m kamel, Study Chair — Alexandria University

IPD SHARING:
Plan to Share IPD: No